CLINICAL TRIAL: NCT06221566
Title: Effectiveness of Muscle Energy Technique (MET) Versus Stretching Exercises In Acute And Subacute Postural Neck Pain. A Randomized Controlled Trial
Brief Title: Effectiveness of Muscle Energy Technique (MET) Versus Stretching Exercises In Acute And Subacute Postural Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NNaqi
Record Dates: First submitted 2024-01-06; First posted 2024-01-24 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2023-12

CONDITIONS: Cervical Pain
Keywords: Proprioceptive Neuromuscular Facilitation (PNF); Static stretching exercises; Visual analog scale
MeSH Terms: conditions — Neck Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Muscle energy technique (MET)
  Interventions: Other: Muscle Energy Technique
- Group B (Active Comparator): Stretching exercise program
  Interventions: Other: Stretching Exercises

INTERVENTIONS:
Other: Muscle Energy Technique — Muscle energy technique (MET) for upper trapezius and levetor scapulae muscle of neck with 7 to 10 second hold, 3 to 5 repetitions.
  Transcutaneous electrical nerve stimulation (TENS) with Cold pack.
  Home exercise program (HEP) will receive by both the groups which will be not supervised by the principal investigator or any other investigator.
  Arms: Group A
Other: Stretching Exercises — Stretching exercises program for upper trapezius and levetor scapulae muscle of neck with 10 second hold, 15 repetitions.
  Transcutaneous electrical nerve stimulation (TENS) with Cold pack.
  Home exercise program (HEP) will receive by both the groups which will be not supervised by the principal investigator or any other investigator.
  Arms: Group B

SUMMARY:
This study will provide better evidence that which technique is more effective in acute and subacute postural neck pain. To find out the effectiveness of Muscle energy technique (MET) and stretching exercises in acute and subacute postural neck pain.

DETAILED DESCRIPTION:
Study Design: Randomized Controlled Trial Study Setting: The study will be conducted at the Institute of Physical Medicine and Rehabilitation, Dow University of Health Sciences, Karachi, Pakistan.

Intervention: This study will identify effects of two intervention approaches. The Experimental group consists of muscle energy technique (MET) for upper trapezius and levetor scapulae muscle of neck. The Control group will receive a stretching exercises program for upper trapezius and levetor scapulae muscle of neck.

ELIGIBILITY:
Inclusion Criteria:

* Targeted population: Students of MBBS, Pharmacy and Doctor of physical therapy.
* Age between 18 and 30 years
* Patient having acute or subacute postural neck pain
* Acute postural neck pain should not last longer than 4weeks
* Subacute postural neck pain should not last longer than 4-12 weeks.

Exclusion Criteria:

* Cervicogenic headaches
* Musculoskeletal disorders involve the nerve root compression, i.e.; (Intervertebral disc dysfunction and derangement syndrome)
* Whiplash associated disorders
* Fibromyalgia
* Spinal cord injury
* Neurological disorders i.e.; (Multiple sclerosis, Young Parkinsonism etc.)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-07-13 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 03 weeks (1st, 8th, 15th, 21st day)
  The pain intensity is measured subjectively on a scale of 0 to 10 cm, where '0 cm' indicates the absence of pain and '10 cm' signifies excruciating pain. Increasing in score suggests worst pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: NIDA NAQI, MSAPT, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Nida Naqi, Karachi, Sindh, Pakistan

REFERENCES:
- [Result] Downie WW, Leatham PA, Rhind VM, Wright V, Branco JA, Anderson JA. Studies with pain rating scales. Ann Rheum Dis. 1978 Aug;37(4):378-81. doi: 10.1136/ard.37.4.378. PMID 686873
- [Result] Hoy DG, Protani M, De R, Buchbinder R. The epidemiology of neck pain. Best Pract Res Clin Rheumatol. 2010 Dec;24(6):783-92. doi: 10.1016/j.berh.2011.01.019. PMID 21665126